CLINICAL TRIAL: NCT03515980
Title: A Phase 1, Open-Label, Parallel Group, Single-Dose Study to Evaluate the Pharmacokinetics, Safety, and Tolerability of BMS-986231 in Participants With Varying Degrees of Hepatic Impairment
Brief Title: An Investigational Study of Experimental Medication BMS-986231 Given in Participants With Different Levels of Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV013-026; 2017-004914-24 (EudraCT Number)
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Liver Dysfunction; Liver Insufficiency; Hepatic Failure; Myocardial Failure; Cardiac Failure; Congestive Heart Failure; Heart Decompensation
MeSH Terms: conditions — Liver Diseases; Hepatic Insufficiency; Liver Failure; Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Mild hepatic impairment (Experimental): Based on Hepatic Function Impairment - Child-Pugh A score 5 to 6 points
  Interventions: Drug: BMS-986231
- Moderate hepatic impairment (Experimental): Based on Hepatic Function Impairment - Child-Pugh B score 7 to 9 points
  Interventions: Drug: BMS-986231
- Severe hepatic impairment (Experimental): Based on Hepatic Function Impairment - Child-Pugh C score 10 to 15 points
  Interventions: Drug: BMS-986231
- Normal hepatic function (Experimental): Based on Hepatic Function Impairment as defined by the investigator
  Interventions: Drug: BMS-986231

INTERVENTIONS:
Drug: BMS-986231 — Intravenous (IV) administration

SUMMARY:
This is an investigational study of experimental Medication BMS-986231 given to participants with weakened or damaged liver function.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Body weight ≥ 45 kg and ≤ 120 kg and BMI ≥ 18 kg/m2 and ≤ 35 kg/m2
* Heart rate ≥ 50 bpm and < 95 bpm
* Women of childbearing potential must have a negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study treatment

Exclusion Criteria:

* Clinically relevant abnormal medical history, abnormal findings on physical examination, vital signs, ECG, or laboratory tests at Screening that the investigator judges as likely to interfere with the objectives of the trial or the safety of the volunteer
* History of chronic headaches (defined as occurring 15 days or more a month, over the previous 3 months), headaches related to caffeine withdrawal (ie, coffee, soda, tea, energy drinks, etc.), or moderately severe to severe headaches
* History of migraine or cluster headaches

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 extrapolated to infinity [AUC(INF)] derived from plasma concentration | Up to 2 days
AUC from time 0 up to time T, where T is the last time point with concentrations above the lower limit of quantitation [AUC(0-T)] derived from plasma concentration | Up to 2 days
Maximum plasma concentration (Cmax) | Up to 2 days

SECONDARY OUTCOMES:
Incidence of adverse events (AE) | Up to 33 days
Incidence of serious adverse events (SAE) | Up to 33 days
Incidence of Laboratory Test Result Abnormalities | Up to 11 days
Clearance (CL) derived from plasma concentration | Up to 2 days
Terminal elimination half-life (t1/2) derived from plasma concentration | Up to 2 days
Time of maximum observed plasma concentration (Tmax) | Up to 2 days
Terminal elimination phase rate constant (λz) derived from plasma concentration | Up to 2 days
Volume of distribution during terminal phase (Vz) derived from plasma concentration | Up to 2 days
Metabolite ratio determined using AUC(INF) for metabolite/AUC(INF) for BMS-986231 [MRAUC(INF)] derived from plasma concentration | Up to 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (4):
- Hungary (2):
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Budapest
  - Clinical Research Unit Hungary, Miskolc
- Poland (2):
  - BioVirtus Centrum Medyczne, Józefów
  - KO-MED Centra Kliniczne Lublin, Lublin

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm